CLINICAL TRIAL: NCT06136078
Title: Appropriateness of MHS Inter-facility Transfers of Traumatic Intracranial Subarachnoid Hemorrhage and Spontaneous Bleeds for Level-1 Advanced Surgical Intervention
Brief Title: Appropriateness of Methodist Health System(MHS) Inter-facility Transfers of Traumatic Intracranial Subarachnoid Hemorrhage and Spontaneous Bleeds for Level-1 Advanced Surgical Intervention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 101.MBSI.2022.A
Record Dates: First submitted 2023-10-18; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Traumatic Intracranial Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: rate of appropriate and inappropriate transfers from Methodist interfacility transfers — Evaluating rate for patients experiencing traumatic intracranial subarachnoid hemorrhage or spontaneous bleeds

SUMMARY:
Brain injuries are common and challenging problems faced by emergency physicians. These diagnoses may include traumatic intracerebral hemorrhage, subarachnoid hemorrhage, ruptured cerebral aneurysms, unruptured cerebral aneurysms, and arteriovenous malformations, which require neurological, neurosurgical, and/or endovascular treatment.

DETAILED DESCRIPTION:
Brain injuries are common and challenging problems faced by emergency physicians. These diagnoses may include traumatic intracerebral hemorrhage, subarachnoid hemorrhage, ruptured cerebral aneurysms, unruptured cerebral aneurysms, and arteriovenous malformations, which require neurological, neurosurgical, and/or endovascular treatment. Depending on the indication and its severity, transfer to a comprehensive stroke center for access to advanced neuro-critical care may be necessary. Comprehensive stroke centers are widely supported and have the resources and infrastructure to have in-house expert stroke providers, teams, operating rooms, and interventional radiology suites that are always available.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Diagnosed with traumatic intracranial subarachnoid hemorrhage or a spontaneous bleed
* Patients originating at Methodist Mansfield medical center (MMMC) or Methodist Charlton medical center(MCMC)and subsequently transferred to Methodist Dallas medical center (MDMC)

Exclusion Criteria:

* Does not meet inclusion criteria defined in section 3.1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Methodist Mansfield Medical Center and Methodist Charlton Medical Center to Methodist Dallas Medical Center for patients experiencing traumatic intracranial subarachnoid hemorrhage or spontaneous bleeds
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
To determine the historical rate of appropriate and inappropriate Methodist interfacility transfers for patients experiencing traumatic intracranial subarachnoid hemorrhage or spontaneous bleed. | 3 days
  Implementation of screening protocols and standardization for interfacility transfers may help to reduce the incidence of unnecessary transfers.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Meyrat, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Clinical Research Institute at Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 2 years

REFERENCES:
- [Background] Alan N, Kim S, Agarwal N, Clarke J, Yealy DM, Cohen-Gadol AA, Sekula RF. Inter-facility transfer of patients with traumatic intracranial hemorrhage and GCS 14-15: The pilot study of a screening protocol by neurosurgeon to avoid unnecessary transfers. J Clin Neurosci. 2020 Nov;81:246-251. doi: 10.1016/j.jocn.2020.09.050. Epub 2020 Oct 15. PMID 33222924